CLINICAL TRIAL: NCT03414307
Title: ROSA Stereotactic Robot-assisted Intracerebral Hemorrhage Clot Evacuation
Brief Title: Stereotactic, Robot-assisted Intracerebral Hemorrhage Clot Evacuation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 Pandemic
Sponsor: Zimmer Biomet (Industry)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0717-1
Record Dates: First submitted 2018-01-16; First posted 2018-01-29 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Intracerebral Hematoma
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Subject enrolled serve as their own control to evaluate the effect of ROSA robotic-assisted intracerebral catheter placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intracerebral hemorrhage (Experimental): Patients with ICH meeting inclusion/exclusion criteria undergo ROSA stereotactic robot-assisted intracerebral catheter placement to evacuate intracerebral or intracranial hemorrhage
  Interventions: Procedure: Intracerebral catheter placement; Device: Robot-assisted intracerebral catheter

INTERVENTIONS:
Procedure: Intracerebral catheter placement — Image guided stereotactic placement of intra-hemorrhage catheters to evacuate intra-cerebral hemorrhage
  Other Names: Stereotactic catheter placement
Device: Robot-assisted intracerebral catheter — ROSA is a robotic device with trajectory planning software that can be used to aid in planning multiple trajectories to large, irregular clots, and aids in navigating into and out of the cerebral hematoma with minimum human error.
  Other Names: ROSA

SUMMARY:
Non-traumatic intracerebral hemorrhage (ICH) affects approximately 100,000 Americans yearly. Up to 30-50% of ICH is fatal, and those patients who survive are often left with significant neurologic dysfunction. In the past, medical management (e.g., control of hypertension, reversal of antiplatelet or anticoagulants) had been the most effective treatment for these patients, given the morbidity and mortality associated with open surgical treatment for evacuation of ICH. However, recent trials have demonstrated that minimally invasive stereotactic neurosurgical procedures to evacuate ICH are safe and result in improved outcomes for these patients.

Initial attempts to evaluate the efficacy of surgical evacuation of ICH found no significant difference between medical management and standard craniotomy for surgical evacuation. Indeed, open surgery was often discouraged for these patients due to the significant morbidity and mortality associated with the surgical procedure itself. However, research has demonstrated that minimally invasive, image guided stereotactic frame-based and frameless methods are effective and safe for the placement of catheters for clot aspiration and fibrinolytic therapy of ICH in the basal ganglia and other deep seated regions. Larger randomized controlled trials have demonstrated that these minimally invasive approaches also offer clinical benefit for these patients.

DETAILED DESCRIPTION:
The introduction of the ROSA stereotactic robot offers an image guided stereotactic approach with greater precision and accuracy than traditional frame-based and frameless methods. While the ROSA has never been used for the placement of intra-hemorrhage catheters, prior applications such as brain biopsies and abscess drainage represent similar surgical procedures which require the same planning, precision, and surgical technique. At the very least, ROSA offers an accurate image guided approach to deep lesions that should be comparable to competitive image guided platforms. At best, ROSA offers superior trajectory planning software, greater ease in planning multiple trajectories to large, irregular clots, and the potential for robot aided navigation into and out of the hematoma which is the greatest source of human error in these cases. For instance, the procedure often requires advancement of a larger aspiration catheter, slow aspiration as the catheter is withdrawn, and then re-advancement of a smaller catheter into the hematoma, which is left in place. The ability to advance and remove catheters in a fixed trajectory with robotic assistance may represent the greatest advantage of ROSA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Head CT demonstrates an acute, spontaneous, supratentorial, primary ICH
* ICH volume ≥30 cc
* Surgery initiated within 48 hours of hospital admission

Exclusion Criteria:

* Pregnancy at the time of surgery
* Underlying vascular lesion defined as causative source of ICH
* Irreversible coagulopathy
* Profound neurological deficit defined as fixed/dilated pupils, bilateral extensor motor posturing
* Infratentorial or brainstem ICH
* Known life expectancy <6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Hematoma volume reduction | Day 1 to Day 4 post operative
  Percentage of hematoma evacuation identified by CT scan

SECONDARY OUTCOMES:
Linear measurement of accuracy | Day 0
  Accuracy of catheter placement is assessed by comparing planned stereotactic trajectories to actual location of the intracerebral catheter. Measure of linear displacement is given in millimeters.
Functional Outcomes measured by modified Rankin Scale (mRS) for neurologic disabilities | Baseline, 3-month, 6-month and 1-year post-operative
  mRS evaluates in a scale 0-6 the degree of disability in patients who have suffered a cerebral stroke or hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Gonzalez, MD, DNP, Study Chair — Zimmer Biomet
Locations (1):
- UPMC Stroke Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hanley DF, Thompson RE, Muschelli J, Rosenblum M, McBee N, Lane K, Bistran-Hall AJ, Mayo SW, Keyl P, Gandhi D, Morgan TC, Ullman N, Mould WA, Carhuapoma JR, Kase C, Ziai W, Thompson CB, Yenokyan G, Huang E, Broaddus WC, Graham RS, Aldrich EF, Dodd R, Wijman C, Caron JL, Huang J, Camarata P, Mendelow AD, Gregson B, Janis S, Vespa P, Martin N, Awad I, Zuccarello M; MISTIE Investigators. Safety and efficacy of minimally invasive surgery plus alteplase in intracerebral haemorrhage evacuation (MISTIE): a randomised, controlled, open-label, phase 2 trial. Lancet Neurol. 2016 Nov;15(12):1228-1237. doi: 10.1016/S1474-4422(16)30234-4. Epub 2016 Oct 11. PMID 27751554
- [Result] Vespa P, Hanley D, Betz J, Hoffer A, Engh J, Carter R, Nakaji P, Ogilvy C, Jallo J, Selman W, Bistran-Hall A, Lane K, McBee N, Saver J, Thompson RE, Martin N; ICES Investigators. ICES (Intraoperative Stereotactic Computed Tomography-Guided Endoscopic Surgery) for Brain Hemorrhage: A Multicenter Randomized Controlled Trial. Stroke. 2016 Nov;47(11):2749-2755. doi: 10.1161/STROKEAHA.116.013837. Epub 2016 Oct 6. PMID 27758940
- [Result] Mendelow AD, Gregson BA, Rowan EN, Murray GD, Gholkar A, Mitchell PM; STICH II Investigators. Early surgery versus initial conservative treatment in patients with spontaneous supratentorial lobar intracerebral haematomas (STICH II): a randomised trial. Lancet. 2013 Aug 3;382(9890):397-408. doi: 10.1016/S0140-6736(13)60986-1. Epub 2013 May 29. PMID 23726393
- [Result] Kim IS, Son BC, Lee SW, Sung JH, Hong JT. Comparison of frame-based and frameless stereotactic hematoma puncture and subsequent fibrinolytic therapy for the treatment of supratentorial deep seated spontaneous intracerebral hemorrhage. Minim Invasive Neurosurg. 2007 Apr;50(2):86-90. doi: 10.1055/s-2007-982503. PMID 17674294